CLINICAL TRIAL: NCT03473145
Title: Sedentary Behavior Interrupted: A Randomized Trial of 3-month Effects on Biomarkers of Healthy Aging and Physical Functioning in the Real World (Project 2)
Brief Title: Sedentary Behavior Interrupted Randomized Controlled Trial (P2)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Sheri Hartman, Assistant Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1P01AG052352-01A1 (NIH)
Record Dates: First submitted 2018-03-14; First posted 2018-03-22 (Actual); Results first posted 2025-11-03 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-09

CONDITIONS: Sedentary Lifestyle
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Health Living Attention Control (Active Comparator): Participants in the attention control condition will receive a healthy aging educational intervention. This group will receive one in-person health coaching sessions and 6 phone counseling sessions.
  Interventions: Behavioral: Health Coaching
- Reduce Sitting (Experimental): Participants in the Reduce Sitting condition will receive an intervention aimed at reducing daily sitting time. This group will receive five in-person health coaching sessions and two phone counseling sessions.
  Interventions: Behavioral: Health Coaching; Device: activPAL inclinometer; Other: Tools to Prompt Standing or Prompt Sit-to-Stand Transitions.
- Sit-to-Stand Transition (Experimental): Participants in the Sit-to-Stand Transition condition will receive an intervention aimed at increasing the daily number of brief sit-to-stand transitions. This group will receive five in-person health coaching sessions and two phone counseling sessions.
  Interventions: Behavioral: Health Coaching; Device: activPAL inclinometer; Other: Tools to Prompt Standing or Prompt Sit-to-Stand Transitions.

INTERVENTIONS:
Behavioral: Health Coaching — Health Coaching sessions will be aimed at goal setting, implementing strategies, overcoming barriers, & relapse prevention.
Device: activPAL inclinometer — Participants in the intervention study arms (B & C) will wear the ActivPAL device for the first 4 weeks of the program and then again in weeks 8 and 9. The device will monitor their sitting and standing time and will allow Health Coaches to provide feedback and will assist the participant in developing an action plan.
  Arms: Reduce Sitting; Sit-to-Stand Transition
Other: Tools to Prompt Standing or Prompt Sit-to-Stand Transitions. — Participants in the intervention study arms (B & C) will receive tools to prompt standing or sit-to-stand transitions such as wearable wrist devices, standing desks or tables (Group B only), mechanical and/or electronic timers, or access to mobile apps or computer programs.
  Arms: Reduce Sitting; Sit-to-Stand Transition

SUMMARY:
Epidemiological findings indicate that older adults do not meet physical activity (PA) guidelines & spend up to 11 hrs/day sitting. Given the high prevalence of sedentary behavior (SB), the higher chronic disease risk in this population, & the age-associated challenges of meeting traditional PA guidelines, involving longer bouts of moderate PA, the investigators hypothesize that older adult health will benefit from new strategies to interrupt sitting. This protocol "Sedentary Behavior Interrupted: A randomized trial of 3-month effects on biomarkers of healthy aging and physical functioning in the real world (Project 2)" is part of a National Institutes of Aging Program Grant called "Sedentary Time & Aging Mortality and Physical Function (STAR). The overall purpose of the STAR program to is to better understand how to interrupt sitting time and the consequences for healthy aging in postmenopausal women. This protocol (also referred to Project 2 of the STAR program) is a 3-arm randomized control trial designed to assess ways of interrupting sitting in 405 overweight, postmenopausal women.

DETAILED DESCRIPTION:
Primary Aims:

In our primary biomarker outcomes of glucose regulation (fasting insulin & glucose, HbA1c, HOMA-IR) & blood pressure (BP):

1. Investigate the 12 week effects of increased standing and additional brief sit-to-stand compared to attention controls.
2. Investigate the dose-response effects of behavioral change on the biomarkers & BP.

Secondary aims

1. Assess the effect of changes in standing and sit-to-stand transitions at 12 weeks on physical, emotional & cognitive functioning.
2. Assess the effect of changes in standing and sit-to-stand transitions at 12 weeks on in vivo skeletal muscle mitochondrial function.

Exploratory aims

1. Explore the possible modifying effect of age on the relationship between intervention conditions & primary & secondary outcomes.
2. Explore the psychosocial & environmental mediators & moderators of changes in sitting time, standing time, and transitions.
3. Explore differences in outcomes between the 2 sitting interruption conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Female;
2. 55 years of age and above;
3. any ethnicity or race;
4. screened to sit for 7 or more hours per day, perform less than 70 sit-to-stand transitions per day
5. ambulatory;
6. medically stable without any health conditions that would inhibit standing or PA;
7. able to give informed consent & comply with study protocols;
8. able to read and write fluently in English;
9. able to travel to study visits; and
10. no menstruation for at least one year;
11. BMI 25-45
12. able to walk, stand and transition without high risk of falling.

Exclusion Criteria:

1. Male;
2. younger than 55 years of age;
3. sit for less than 7 hours per day, perform 71 or more sit-to-stand transitions per day
4. mental state that would preclude complete understanding of the protocol or compliance;
5. physical limitations to completing any of the study conditions;
6. menstruation less than one year prior;
7. unable to complete the Short Physical Performance Battery,
8. Active cancer
9. body Mass Index <25 or >45kg/m2,
10. use of insulin

Min Age: 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 407 (Actual)
Dates: Start 2018-05-30 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UC San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hartman SJ, LaCroix AZ, Sears DD, Natarajan L, Zablocki RW, Chen R, Patterson JS, Dillon L, Sallis JF, Schenk S, Dunstan DW, Owen N, Rosenberg DE. Impacts of Reducing Sitting Time or Increasing Sit-to-Stand Transitions on Blood Pressure and Glucose Regulation in Postmenopausal Women: Three-Arm Randomized Controlled Trial. Circulation. 2025 Aug 26;152(8):492-504. doi: 10.1161/CIRCULATIONAHA.124.073385. Epub 2025 Jul 25. PMID 40709462
- [Derived] Zablocki RW, Hartman SJ, Di C, Zou J, Carlson JA, Hibbing PR, Rosenberg DE, Greenwood-Hickman MA, Dillon L, LaCroix AZ, Natarajan L. Using functional principal component analysis (FPCA) to quantify sitting patterns derived from wearable sensors. Int J Behav Nutr Phys Act. 2024 Apr 26;21(1):48. doi: 10.1186/s12966-024-01585-8. PMID 38671485
- [Derived] Hartman SJ, Dillon LW, LaCroix AZ, Natarajan L, Sears DD, Owen N, Dunstan DW, Sallis JF, Schenk S, Allison M, Takemoto M, Herweck AM, Nguyen B, Rosenberg DE. Interrupting Sitting Time in Postmenopausal Women: Protocol for the Rise for Health Randomized Controlled Trial. JMIR Res Protoc. 2021 May 13;10(5):e28684. doi: 10.2196/28684. PMID 33983131

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Health Living Attention Control | Reduce Sitting | Sit-to-Stand Transition
Started | 135 | 136 | 136
Completed | 130 | 130 | 128
Not Completed | 5 | 6 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Health Living Attention Control | Reduce Sitting | Sit-to-Stand Transition | Total
Number analyzed (Participants) | 135 | 136 | 136 | 407
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.76 (7.43) | 68.39 (4.66) | 67.29 (6.55) | 67.81 (32.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 135 | 136 | 136 | 407
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 13 | 10 | 35
  Not Hispanic or Latino | 123 | 123 | 124 | 370
  Unknown or Not Reported | 0 | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1 | 2
  Asian | 3 | 2 | 5 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 7 | 4 | 4 | 15
  White | 120 | 126 | 125 | 371
  More than one race | 2 | 2 | 1 | 5
  Unknown or Not Reported | 2 | 2 | 0 | 4
Region of Enrollment [Number; unit: participants]
  United States | 135 | 136 | 136 | 407

OUTCOME MEASURES:

1. Primary Outcome: Insulin Regulation (mU/L)
Description: Mean Insulin (mU/L) collected via fasting blood draw at Baseline and 3-Months
Time Frame: 3 months
Measure: Mean (95% Confidence Interval); unit: mU/L
Arm/Group | Health Living Attention Control | Reduce Sitting | Sit-to-Stand Transition
Number analyzed (Participants) | 131 | 133 | 135
mU/L
  Baseline Mean | 15.93 [14.25 to 17.62] | 15.68 [14.03 to 17.33] | 15.27 [13.68 to 16.86]
  3-Month Mean | 16.72 [14.94 to 18.51] | 15.85 [14.17 to 17.53] | 14.84 [13.26 to 16.41]

2. Secondary Outcome: Self-Reported Physical Functioning
Description: Self-reported physical functioning was assessed using the Rand SF 36-Item Health Survey that assesses 8 health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. The range of scores is 0 - 100 with higher scores meaning better physical functioning.
Time Frame: 3 months
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Health Living Attention Control | Reduce Sitting | Sit-to-Stand Transition
Number analyzed (Participants) | 135 | 136 | 136
score on a scale
  Baseline Mean | 74.9 (1.81) | 72.8 (1.81) | 75.8 (1.81)
  3-Months Mean | 75.9 (1.83) | 74.6 (1.83) | 80.5 (1.84)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected while the participants were active in the study for 3-months.
Arm/Group | Health Living Attention Control | Reduce Sitting | Sit-to-Stand Transition
All-Cause Mortality (participants affected / at risk) | 0/135 | 0/136 | 0/136
Serious Adverse Events (participants affected / at risk) | 0/135 | 0/136 | 0/136
Other Adverse Events (participants affected / at risk) | 8/135 | 28/136 | 26/136
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Health Living Attention Control (N=135) | Reduce Sitting (N=136) | Sit-to-Stand Transition (N=136)
Skin Irritation (Skin and subcutaneous tissue disorders) | 8 (9) | 16 (16) | 18 (18) — Skin Irritation from wearing the study devices
Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 12 (12) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-05-01): https://cdn.clinicaltrials.gov/large-docs/45/NCT03473145/Prot_001.pdf
  • Statistical Analysis Plan (2025-08-26): https://cdn.clinicaltrials.gov/large-docs/45/NCT03473145/SAP_002.pdf
  • Informed Consent Form (2022-03-29): https://cdn.clinicaltrials.gov/large-docs/45/NCT03473145/ICF_000.pdf